CLINICAL TRIAL: NCT05954884
Title: Community-based HEARTS Intervention (Pilot)
Acronym: CB-HEARTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Heart Foundation of Bangladesh (Other)
Collaborators: National Heart Foundation Hospital and Research Institute (Unknown); Johns Hopkins University (Other); Non-communicable Disease Control Programme, Directorate General of Health Services, Bangladesh (Unknown); Community Based Health Care, Directorate General of Health Services, Bangladesh (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BMRC/NREC/2022-2025/102
Record Dates: First submitted 2023-07-13; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): This is a single-arm pilot study and all participants will receive the intervention. Participants will be diagnosed and treated for hypertension at Community Clinic (CC) by a Community Health Care Provider (CHCP) under telemedicine supervision from a Medical Officer at the Upazila Health Complex (UHC).
  Interventions: Other: Telemedicine-based WHO HEARTS package

INTERVENTIONS:
Other: Telemedicine-based WHO HEARTS package — Interventions in this study will include-
  1. Community- and team-based model of hypertension care delivery
  2. Opportunistic hypertension screening at Community Clinic (CC) by Community Health Care Provider (CHCP)
  3. Use of a hypertension treatment protocol with amlodipine and losartan and standardized approach to measuring and monitoring BP, retaining participants in care, and promoting adherence
  4. Use of Simple App to document BP readings and medications/dosage and to monitor hypertension care delivery at the CC through utilities including dashboards
  5. Establishment of telemedicine service between CC and Upazila Health Complex (UHC)
  6. Community-based, multi-month prescription refills from CC
  7. Training of clinic and research staff on BP measurement following standard techniques
  8. Site monitoring and mentorship to ensure screening and patient enrollment/registration
  9. Use of text messages to promote follow-up visits and medication adherence

SUMMARY:
The goal of this pilot study is to assess the feasibility of health system change intervention with a focus on recruitment of patients with hypertension, initiation of antihypertensive medication, and retention of patients in care at the Community Clinics (CC) with a goal of finalizing the key features of a team- and community-based intervention in rural Bangladesh.

Patients with uncomplicated hypertension will be enrolled, their medical treatment will be provided from CC by a Community Health Care Provider (CHCP) according to the telemedicine-based instruction of Medical Officer from Upazila Health Complex (UHC) with provision of referral to UHC for an in-person evaluation. Participants will be followed up periodically and their medicine will be refilled accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Patients residing in the catchment area of the selected 4 Community Clinics under selected 2 Upazila Health Complexes (UHCs)
* Aged 18 years and older
* Raised BP during screening [Systolic BP ≥140 mmHg and/or diastolic BP ≥90 mmHg (based on an average of minimum two measurements)]
* Not currently taking antihypertensive medications
* Eligible for the HEARTS technical package, defined as not being treated for an acute illness or medical emergency and not having a terminal illness

Exclusion Criteria:

* Patients with cardiovascular diseases, chronic kidney diseases (as evident by previous laboratory report of serum creatinine or urinary protein more than ++ on dipstick test prior to the enrollment), diabetes, or BP >180/110 mmHg (based on the mean of last two BP measurements) at screening or after 14 days of recommended lifestyle modification will be excluded and referred directly to UHC for further management
* Pregnancy or intent to become pregnant
* Patients who otherwise meet inclusion criteria but decline to participate in the hypertension program evaluation or do not provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Enrollment proportion | 6 months from enrollment
  The proportion of eligible individuals with raised BP identified at the Community Clinic (CC) who were enrolled, defined as those started on meds within 6 months of diagnosis
Short-term, intermediate, and long-term retention in care | 3 months from enrollment for short-term retention in care, 6 to 12 months for intermediate retention in care, and 12 to 18 months for long-term retention in care
  The proportion of enrolled individuals with raised BP who had a follow-up visit within 3 months of enrollment (short-term retention in care), between 6 and 12 months (intermediate retention in care), and between 12 and 18 months (long-term retention in care)

SECONDARY OUTCOMES:
Blood pressure control | 3, 6, 12, and 18 months from enrollment
  The proportion of those enrolled at the Community Clinic with BP controlled (<140/90 mmHg) at 3, 6, 12, and 18 months (denominator includes patients who do not return for follow up BP measurement)

CONTACTS AND LOCATIONS:
Overall Officials: Sohel R Choudhury, PhD, Principal Investigator — National Heart Foundation Hospital and Research Institute